CLINICAL TRIAL: NCT07230834
Title: A Phase 1 Dose-Escalation and Repeated-Dose Study of the Safety and Tolerability of Intravitreal Pozelimab in Participants With Geographic Atrophy
Brief Title: Intravitreal (IVT) Pozelimab for Geographic Atrophy (GA) in Adult Participants
Acronym: VIENNA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3918-AMD-2501; 2025-521758-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Geographic Atrophy (GA)
Keywords: Age-related Macular Degeneration (AMD); GA secondary to AMD
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A will not be masked (Open label) and part B is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental)
  Interventions: Drug: Pozelimab
- Part B (Experimental)
  Interventions: Drug: Pozelimab

INTERVENTIONS:
Drug: Pozelimab — Administered per the protocol
  Other Names: REGN3918

SUMMARY:
This study is researching an experimental drug called pozelimab (called "study drug"). The study is focused on people with a condition where certain parts of the eye's retina stop working over time, which can make it harder to see. This is called geographic atrophy (GA).

The aim of the study is to see how safe and tolerable the study drug is when used as an injection in the eye.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood and the fluid in the eye at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Study eye with diagnosis of GA of the macula secondary to AMD, as determined by the investigator
2. Study eye with total GA area measuring approximately one disc area or greater in size (2.5 mm^2 or larger) at screening, as determined by the Central Reading Center (CRC), as described in the protocol
3. Best-Corrected Visual Acuity (BCVA) of 60 letters or worse using the Early Treatment Diabetic Retinopathy Score (ETDRS) charts (Snellen equivalent of ~ ≤20/63) in the study eye at screening and baseline visit

Key Exclusion Criteria:

1. GA (macular atrophy) in either eye due to causes other than dry AMD
2. History or current evidence of macular neovascularization and/or retinal exudation in either eye
3. Concurrent eye disease (elevated Intraocular Pressure (IOP) >25mm Hg, diabetic retinopathy, ocular infections/inflammation)
4. Prior or current intravitreal (IVT) treatment of any kind for any indication in either the study or fellow eye, except complement inhibitor therapy for GA, as long as last dose was ≥3 months prior to screening
5. Any prior systemic treatment for dry AMD, except oral supplements or vitamins
6. History or current use of systemic complement inhibitor therapy

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2028-07-03 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of ocular Treatment-Emergent Adverse Event (TEAEs) in the study eye | Through week 8
  Part A
Occurrence of ocular TEAEs in the study eye | Through week 16
  Part B
Occurrence of systemic TEAEs | Through week 8
  Part A
Occurrence of systemic TEAEs | Through week 16
  Part B

SECONDARY OUTCOMES:
Concentrations of pozelimab in serum | Through week 8
  Part A
Concentrations of pozelimab in serum | Through week 16
  Part B
Occurrence of Anti-Drug Antibody (ADA) to pozelimab | Through week 8
  Part A
Magnitude of ADA to pozelimab | Through week 8
  Part A
Occurrence of ADA to pozelimab | Through week 16
  Part B
Magnitude of ADA to pozelimab | Through week 16
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Colorado Retina Associates, Lakewood, Colorado
  - Austin Retina Associates, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/